CLINICAL TRIAL: NCT00035633
Title: A Phase III Study of Entecavir vs Lamivudine in Adults With Chronic Hepatitis B Infection and Positive for Hepatitis B E Antigen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: AI463-022
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

INTERVENTIONS:
Drug: Entecavir

SUMMARY:
The purpose of this clinical research study is to assess the safety effectiveness of entecavir, as compared to lamivudine, in the treatment of adults with chronic hepatitis B infection who are hepatitis B e antigen positive.

ELIGIBILITY:
* Male and female subjects =/> 16 years of age (or minimum age required in a given country) with history of chronic hepatitis B infection;
* Documentation of positive Hepatitis B e antigen (HBeAg) status.;
* The absence of coinfection with immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV);
* The absence of other forms of liver disease e.g., alcoholic, autoimmune, biliary disease;
* Less than 12 weeks prior therapy with nucleoside or nucleotide analogue antiviral agents with activity against hepatitis B (e.g., adefovir, famciclovir and lamivudine)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Local Investigator, Birmingham, Alabama
  - Local Investigator, Tucson, Arizona
  - Local Investigator, La Jolla, California
  - Local Investigator, Los Angeles, California
  - Local Investigator, Orange, California
  - Local Investigator, Palo Alto, California
  - Local Institution, San Francisco, California
  - Local Investigator, Torrance, California
  - Local Investigator, Farmington, Connecticut
  - Local Investigator, Miami, Florida
  - Local Investigator, Atlanta, Georgia
  - Local Investigator, Honolulu, Hawaii
  - Local Investigator, Chicago, Illinois
  - Local Investigator, Iowa City, Iowa
  - Local Investigator, Boston, Massachusetts
  - Local Investigator, Worcester, Massachusetts
  - Local Investigator, Ann Arbor, Michigan
  - Local Investigator, Royal Oak, Michigan
  - Local Investigator, Saint Paul, Minnesota
  - Local Investigator, Manhasset, New York
  - Local Investigator, New York, New York
  - Local Investigator, Rochester, New York
  - Local Investigator, Charlotte, North Carolina
  - Local Investigator, Cleveland, Ohio
  - Local Investigator, Philadelphia, Pennsylvania
  - Local Investigator, Pittsburgh, Pennsylvania
  - Investigator Meeting, Providence, Rhode Island
  - Local Investigator, Nashville, Tennessee
  - Local Investigator, Dallas, Texas
  - Local Investigator, Fairfax, Virginia
  - Local Investigator, Richmond, Virginia
  - Local Investigator, Seattle, Washington

REFERENCES:
- [Result] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137